CLINICAL TRIAL: NCT00731120
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of 2 Doses of Lu AA21004 in Acute Treatment of Adults With Generalized Anxiety Disorder
Brief Title: Study of Efficacy and Safety of Vortioxetine (Lu AA21004) in Treating Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_309; U1111-1114-2380 (Registry Identifier: WHO)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Mood Disorder; Affective Disorder; Anxiety Disorder; Drug Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Mood Disorders; Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 2.5 mg (Experimental): Vortioxetine 2.5 mg encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate-release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 10 mg; Vortioxetine 2.5 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 2.5 mg and 10 mg vortioxetine, once daily (QD), in adults with generalized anxiety disorder.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned to receive either 2.5 mg or 10 mg of vortioxetine or a placebo once daily for an eight week treatment period.

Participants will be seen weekly during the first 2 weeks of treatment, and then every 2 weeks up to the end of the 8-week treatment period. Total commitment time is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of Generalized Anxiety Disorder according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR®) criteria (classification code 300.02).
* Has a Hamilton Anxiety Scale total score ≥ 20.
* Has a Hamilton Anxiety Scale score ≥ 2 on both item 1 (anxious mood) and item 2 (tension).
* Has a Montgomery-Åsberg Depression Rating Scale total score ≤16.

Exclusion Criteria:

* Has 1 or more of the following:

  * Any current psychiatric disorder other than Generalized Anxiety Disorder as defined in the DSM-IV-TR (as assessed by the Mini International Neuropsychiatric Interview [MINI]).
  * Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR and participant must have a negative urine drug screen prior to Baseline.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc.).
  * Any Axis II disorder that might compromise the study.
* Is taking excluded medications.
* Has a significant risk of suicide according to the investigator's opinion or has a score ≥5 on Item 10 (suicidal thoughts) of the Montgomery-Åsberg Depression Rating Scale or has made a suicide attempt in the previous 6 months.
* Has previously failed to respond to adequate treatment with selective serotonin reuptake inhibitors and/or serotonin-norepinephrine reuptake inhibitors.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a clinically significant unstable illness.
* Has an alanine aminotransferase, aspartate aminotransferase, or total bilirubin level > 1.5 times the upper limit of normal.
* Has a serum creatinine of > 1.5 × the upper limit of normal.
* Has a previous history of cancer that had been in remission for less than 5 years.
* Has thyroid stimulating hormone value outside the normal range.
* Has an abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (40):
- United States (40):
  - Birmingham, Alabama
  - Anaheim, California
  - Cerritos, California
  - Costa Mesa, California
  - Orange, California
  - Redlands, California
  - Cromwell, Connecticut
  - Norwich, Connecticut
  - Hockessin, Delaware
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Lady Lake, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Libertyville, Illinois
  - Valparaiso, Indiana
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Boston, Massachusetts
  - Braintree, Massachusetts
  - Pittsfield, Massachusetts
  - St Louis, Missouri
  - Cherry Hill, New Jersey
  - Fresh Meadows, New York
  - New York, New York
  - Olean, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Emmaus, Pennsylvania
  - Philadelphia, Pennsylvania
  - Reading, Pennsylvania
  - North Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Midlothian, Virginia
  - Waukesha, Wisconsin

REFERENCES:
- [Derived] Mahableshwarkar AR, Jacobsen PL, Serenko M, Chen Y. A randomized, double-blind, fixed-dose study comparing the efficacy and tolerability of vortioxetine 2.5 and 10 mg in acute treatment of adults with generalized anxiety disorder. Hum Psychopharmacol. 2014 Jan;29(1):64-72. doi: 10.1002/hup.2371. PMID 24424707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 41 investigative sites in the United States from 17 June 2008 to 16 February 2009.
Pre-assignment Details: Participants with a diagnosis of generalized anxiety disorder were enrolled equally in one of three treatment groups, once a day placebo or 2.5 or 10 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Started | 153 | 152 | 152
Treated | 153 | 151 | 152
Completed | 111 | 109 | 116
Not Completed | 42 | 43 | 36
Not completed — Adverse Event | 7 | 6 | 8
Not completed — Lack of Efficacy | 4 | 5 | 4
Not completed — Noncompliance with Study Drug | 3 | 3 | 1
Not completed — Protocol Deviations | 1 | 6 | 1
Not completed — Withdrawal of Consent | 13 | 8 | 4
Not completed — Lost to Follow-up | 10 | 15 | 17
Not completed — Other | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg | Total
Number analyzed (Participants) | 153 | 152 | 152 | 457
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.45) | 40.8 (13.81) | 43.3 (14.99) | 41.2 (14.15)
Age, Customized [Number; unit: participants]
  ≤55 years | 136 | 127 | 120 | 383
  >55 years | 17 | 25 | 32 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 103 | 96 | 304
  Male | 48 | 49 | 56 | 153
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 13 | 18 | 15 | 46
  Non-Hispanic/Non-Latino | 140 | 134 | 137 | 411
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 105 | 110 | 112 | 327
  Black | 46 | 38 | 38 | 122
  Asian | 2 | 3 | 2 | 7
  American Indian or Alaska Native | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 153 | 152 | 152 | 457
Weight [Mean (Standard Deviation); unit: kg] | 82.66 (20.731) | 84.48 (22.727) | 85.67 (23.249) | 84.27 (22.245)
Height [Mean (Standard Deviation); unit: cm] | 168.31 (9.994) | 168.63 (8.932) | 168.86 (10.032) | 168.60 (9.649)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.10 (6.595) | 29.69 (7.817) | 30.04 (7.792) | 29.61 (7.415)
Smoking Classification [Number; unit: participants]
  Never Smoked | 87 | 72 | 84 | 243
  Current smoker | 44 | 51 | 46 | 141
  Ex-smoker | 22 | 29 | 22 | 73
Alcohol Consumption [Number; unit: participants]
  Never | 50 | 42 | 44 | 136
  Once monthly or less often | 52 | 54 | 56 | 162
  Once a week | 33 | 28 | 29 | 90
  2 to 6 times per week | 17 | 23 | 22 | 62
  Daily | 1 | 5 | 1 | 7
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a scale | 25.2 (3.86) | 25.0 (3.60) | 24.5 (3.71) | 24.9 (3.73)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.4 (0.54) | 4.3 (0.49) | 4.3 (0.47) | 4.3 (0.50)
Hospital Anxiety and Depression - Anxiety subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 13.9 (3.27) | 13.2 (3.56) | 13.2 (3.17) | 13.4 (3.35)
Hospital Anxiety and Depression - Depression subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Depression sub-scale consists of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). The depression subscale focuses on the state of lost interest and diminished pleasure response. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 8.7 (3.67) | 8.0 (3.80) | 8.0 (3.60) | 8.3 (3.70)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 12.73 (2.417) | 12.64 (2.502) | 13.04 (2.521) | 12.80 (2.481)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Least Squares (LS) means were from an analysis of covariance (ANCOVA) model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: The full analysis set (FAS) included all randomized patients who received at least 1 dose of study drug, and had at least 1 post-baseline value for assessment of primary efficacy. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
scores on a scale | -9.87 (0.584) | -10.75 (0.569) | -10.68 (0.581)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; P-values were tested at the 5% significance level (ie, statistical significance if P<0.05). To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 10 mg and 2.5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.05, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.279, ANCOVA — Hierarchical testing stopped at 10 mg versus placebo for HAM-A total score at Week 8 in the testing sequence, a nominal p-value is provided; Analysis of covariance (ANCOVA), with treatment and center as fixed factors and baseline HAM-A as a covariate; LS Mean Difference = -0.87, 95% CI 2-sided [-2.45 to 0.71], Standard Error of Mean 0.803
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.306, ANCOVA — Pre-specified sequential statistical testing procedure indicates that when p-value >0.05, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; Analysis of covariance (ANCOVA), with treatment and center as fixed factors and baseline HAM-A as a covariate; LS Mean Difference = -0.81, 95% CI 2-sided [-2.36 to 0.74], Standard Error of Mean 0.791

2. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
scores on a scale
  Week 1 (n=147, 142, 143) | -5.07 (0.433) | -5.29 (0.423) | -5.30 (0.433)
  Week 2 (n=148, 144, 146) | -7.41 (0.501) | -8.11 (0.488) | -8.05 (0.499)
  Week 4 (n=148, 144, 146) | -8.88 (0.566) | -9.45 (0.551) | -9.54 (0.564)
  Week 6 (n=148, 144, 146) | -9.54 (0.565) | -10.35 (0.550) | -10.50 (0.563)

3. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Week 8
Description: Response was defined as a participant with a ≥50% decrease from Baseline in the HAM-A total score. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Baseline and Week 8
Population: Full analysis set; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
percentage of participants | 41.9 | 46.5 | 41.8

4. Secondary Outcome: Percentage of Participants in HAM-A Remission at Week 8
Description: Remission is defined as a Hamilton Anxiety Scale (HAM-A) total score ≤ 7. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Week 8
Population: Full analysis set; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
percentage of participants | 21.6 | 21.5 | 19.2

5. Secondary Outcome: Clinical Global Impression Scale-Global Improvement (CGI-I) at Each Week Assessed
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from an ANCOVA model adjusting for Baseline CGI-S score, center, and treatment.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
scores on a scale
  Week 1 (n=146, 141, 143) | 3.35 (0.071) | 3.30 (0.070) | 3.38 (0.071)
  Week 2 (n=148, 143, 146) | 2.99 (0.083) | 2.91 (0.081) | 2.92 (0.083)
  Week 4 (n=148, 144, 146) | 2.87 (0.089) | 2.75 (0.086) | 2.69 (0.088)
  Week 6 (n=148, 144, 146) | 2.68 (0.089) | 2.58 (0.087) | 2.60 (0.088)
  Week 8 (n=148, 144, 146) | 2.60 (0.095) | 2.56 (0.093) | 2.51 (0.095)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness (CGI-S)
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from an ANCOVA model adjusting for Baseline score, center, and treatment.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
scores on a scale
  Week 1 (n=146, 140, 143) | -0.40 (0.054) | -0.47 (0.053) | -0.37 (0.054)
  Week 2 (n=148, 143, 146) | -0.68 (0.072) | -0.82 (0.070) | -0.69 (0.071)
  Week 4 (n=148, 144, 146) | -0.82 (0.081) | -1.01 (0.079) | -0.93 (0.081)
  Week 6 (n=148, 144, 146) | -0.93 (0.083) | -1.14 (0.081) | -1.03 (0.082)
  Week 8 (n=148, 144, 146) | -1.10 (0.090) | -1.21 (0.088) | -1.14 (0.090)

7. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HAD) Scales
Description: The HAD scale is completed by the participant and comprises two subscales, one measuring depression (focusing on the state of lost interest and diminished pleasure response) and one measuring anxiety (including anxious mood, restlessness, anxious thoughts, panic attacks). Each subscale is made up of 7 items that are assessed on a scale of 0 = no anxiety/depression to 3 = severe feeling of anxiety/depression. Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. Scores for the depression and anxiety subscales are summed separately and not combined, with each score ranging from 0 to 21 (maximal severity). LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4 and 8.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
scores on a scale
  Anxiety Scale at Week 1 (n=147, 142, 143) | -1.64 (0.266) | -2.07 (0.258) | -2.03 (0.264)
  Anxiety Scale at Week 4 (n=148, 144, 146) | -2.81 (0.343) | -3.66 (0.333) | -3.39 (0.339)
  Anxiety Scale at Week 8 (n=148, 144, 146) | -3.63 (0.365) | -4.29 (0.354) | -4.20 (0.361)
  Depression Scale at Week 1 (n=147, 142, 143) | -0.71 (0.226) | -1.35 (0.220) | -1.15 (0.225)
  Depression Scale at Week 4 (n=148, 144, 146) | -1.66 (0.272) | -2.23 (0.265) | -2.10 (0.271)
  Depression Scale at Week 8 (n=148, 144, 146) | -1.76 (0.308) | -2.56 (0.300) | -2.21 (0.306)

8. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: Full analysis set with available data at Baseline; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 124 | 113 | 109
scores on a scale | -4.26 (0.617) | -5.73 (0.623) | -5.24 (0.657)

9. Secondary Outcome: Change From Baseline in 36-item Short-form Health Survey (SF-36)
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The 8 health concepts are: 1. Limitation in physical activities because of health problems. 2. Limitations in usual role activities because of physical health problems. 3. Bodily pain. 4. Limitations in social activities because of physical or emotional problems. 5. General mental health (psychological distress and well-being). 6. Limitations in usual role activities because of emotional problems. 7. Vitality (energy and fatigue). 8. General health perception. Each scale ranges from 0 (best) - 100 (worst). LS means were from an ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: Full analysis set with a Baseline SF-36 measurement; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 146 | 141 | 141
scores on a scale
  Physical functioning subscore | 0.46 (1.513) | 2.69 (1.478) | 2.07 (1.517)
  Role - physical subscore | 4.44 (2.018) | 8.17 (1.972) | 6.17 (2.026)
  Bodily pain subscore | 5.90 (1.901) | 10.67 (1.855) | 8.12 (1.905)
  General health subscore | 4.44 (1.289) | 7.01 (1.258) | 5.90 (1.292)
  Vitality subscore | 12.35 (1.782) | 15.62 (1.740) | 14.33 (1.783)
  Social functioning subscore | 15.35 (2.075) | 18.38 (2.025) | 17.56 (2.070)
  Role-emotional subscore | 15.16 (2.076) | 21.72 (2.028) | 16.60 (2.081)
  Mental health subscore | 12.93 (1.642) | 17.25 (1.608) | 14.74 (1.643)

10. Secondary Outcome: Health Care Resource Utilization Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 148 | 144 | 146
participants
  Baseline: Any resource use | 32 | 34 | 32
  Baseline: Any hospitalization-related services | 2 | 1 | 1
  Baseline: Hospitalization related to anxiety | 1 | 0 | 0
  Baseline: Any sick leave | 5 | 13 | 10
  Baseline: Sick leave related to anxiety | 4 | 8 | 4
  Week 8: Any resource use | 14 | 23 | 19
  Week 8: Any hospitalization-related service | 3 | 0 | 1
  Week 8: Hospitalization related to anxiety | 0 | 0 | 0
  Week 8: Any sick leave | 5 | 6 | 8
  Week 8: Sick leave related to anxiety | 1 | 4 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of double-blind study medication through 30 days after permanent discontinuation of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 10 mg
Serious Adverse Events (participants affected / at risk) | 1/153 | 2/151 | 1/152
Other Adverse Events (participants affected / at risk) | 70/153 | 72/151 | 83/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=153) | Vortioxetine 2.5 mg (N=151) | Vortioxetine 10 mg (N=152)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=153) | Vortioxetine 2.5 mg (N=151) | Vortioxetine 10 mg (N=152)
Palpitations (Cardiac disorders) | 1 | 5 | 0
Nausea (Gastrointestinal disorders) | 13 | 24 | 37
Diarrhoea (Gastrointestinal disorders) | 11 | 13 | 17
Dry mouth (Gastrointestinal disorders) | 17 | 14 | 12
Constipation (Gastrointestinal disorders) | 6 | 4 | 9
Vomiting (Gastrointestinal disorders) | 4 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 1
Fatigue (General disorders) | 2 | 3 | 7
Irritability (General disorders) | 2 | 4 | 1
Nasopharyngitis (Infections and infestations) | 8 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 6
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 5
Influenza (Infections and infestations) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 3
Headache (Nervous system disorders) | 17 | 20 | 18
Dizziness (Nervous system disorders) | 6 | 7 | 6
Somnolence (Nervous system disorders) | 6 | 5 | 2
Sedation (Nervous system disorders) | 4 | 5 | 5
Insomnia (Psychiatric disorders) | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.